CLINICAL TRIAL: NCT05967494
Title: Assessing Patient Engagement and Understanding in Chronic Fatigue Syndrome Clinical Trials
Brief Title: Discovering Trends in Chronic Fatigue Syndrome Patients' Clinical Study Experiences
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 84606875
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Fatigue Syndrome
Keywords: Chronic Fatigue Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study seeks to delve into the firsthand experiences of patients diagnosed with chronic fatigue syndrome who partake in a separate clinical trial featuring a specific medical intervention. The primary emphasis will be on meticulously tracking the rates of trial completion and withdrawal among these individuals.

The data collected from this study will help improve future outcomes for all chronic fatigue syndrome patients as well as those in under-represented demographic groups.

ELIGIBILITY:
Inclusion Criteria:

* Signed Written Informed Consent
* Aged ≥ 18 years old
* No prior treatment for chronic fatigue syndrome

Exclusion Criteria:

* Participant is actively receiving study therapy in another
* Inability to provide written informed consent
* Women of childbearing potential without a negative pregnancy test; or women who are lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic fatigue syndrome who are actively considering enrolling in a clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to join in a chronic fatigue syndrome clinical trial | 3 months
Number of chronic fatigue syndrome patients who remain in clinical trial until completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meng XD, Guo HR, Zhang QY, Li X, Chen Y, Li MY, Zhuo XM, Wang MJ, Shan K, Gong YN, Li NC, Chen B, Chen ZL, Guo Y. The effectiveness of cupping therapy on chronic fatigue syndrome: A single-blind randomized controlled trial. Complement Ther Clin Pract. 2020 Aug;40:101210. doi: 10.1016/j.ctcp.2020.101210. Epub 2020 Jun 20. PMID 32891286
- [Background] Kim DY, Lee JS, Park SY, Kim SJ, Son CG. Systematic review of randomized controlled trials for chronic fatigue syndrome/myalgic encephalomyelitis (CFS/ME). J Transl Med. 2020 Jan 6;18(1):7. doi: 10.1186/s12967-019-02196-9. PMID 31906979
- [Background] Galeoto G, Sansoni J, Valenti D, Mollica R, Valente D, Parente M, Servadio A. The effect of physiotherapy on fatigue and physical functioning in chronic fatigue syndrome patients: A systematic review. Clin Ter. 2018 Jul-Aug;169(4):e184-e188. doi: 10.7417/T.2018.2076. PMID 30151552

DOCUMENTS (1):
  • Informed Consent Form (2023-07-21): https://cdn.clinicaltrials.gov/large-docs/94/NCT05967494/ICF_000.pdf